CLINICAL TRIAL: NCT00662480
Title: Randomized Preventive Vascular Screening Trial of 65-74 Year Old Men in the Central Region of Denmark
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Jes S. Lindholt, Vascular Research Unit, Department of Vascular Surgery, Viborg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: M-20080028
Record Dates: First submitted 2008-04-15; First posted 2008-04-21 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Abdominal Aortic Aneurysms; Peripheral Arterial Disease; Hypertension
Keywords: population; screening; abdominal aortic aneurysms; peripheral arterial disease; hypertension; Prevention
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Peripheral Arterial Disease; Hypertension | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Invited to screening for hypertension, lower limb atherosclerosis and abdominal aortic aneurysm
  Interventions: Procedure: Screening for hypertension, lower limb atherosclerosis and abdominal aortic aneurysm
- 2 (No Intervention): Participants which are not offered vascular screening

INTERVENTIONS:
Procedure: Screening for hypertension, lower limb atherosclerosis and abdominal aortic aneurysm — Invited to vascular screening
  Arms: 1

SUMMARY:
Well-documented health benefits may be achieved through prophylactic screening for cardiovascular disease. The advantages are fewer premature deaths and a reduction in the number of hospital admissions and amputations. Furthermore, hospitals will benefit from the derived reduction in the pressure on surgery and intensive care capacities at vascular surgery departments.

It therefore seems extremely relevant to offer joint screening for abdominal aortic aneurysm, peripheral arterial disease and hypertension, even if the benefit and costs of such a measure are not currently known.

Consequently, the primary objective of the study is to establish the effect and cost-efficiency of a joint circulation screening programme for 40,000 men aged 65-74 years in a randomised, clinically controlled study.

The project manager will train six nurses to measure ABI and perform ultrasound scans of the aorta. The nurses form three teams which will each be equipped with a portable Doppler, blood pressure cuff and portable ultrasound scanner. Each team will operate from the hospitals in the Region. Civil registration number (in Danish: CPR), name and address information will be supplied by the Clinical Epidemiological Department (CED), which will also perform the randomisation in groups of approx. 1,000 to avoid too long a period from data extraction to invitation. Half of the randomised subjects will be invited to participate in a circulation examination focused on PAD, AAA and hypertension, while the other half will be controls Men with positive findings are informed and proper preventive actions is taken. Annual controls are offered, and AAA exceeding 5.5 cm in diameter is offered operation.

The primary efficiency variables are death, cardiovascular death and AAA-death. The secondary efficiency variables are hospital services related to cardiovascular conditions and costs for such services in accordance with current DRG rates.

The entire population, the controls as well as the screening group, will be monitored for a period of 10 years. Information concerning deaths, including date of death, is obtained from the Civil Registration System, information on visits to outpatient clinics and hospital admissions caused by cardiovascular conditions including amputations is obtained from the National Patient Registry. From the Danish Causes of Death Registry information on cause of death is collected. The information is classified with regards to cause; AAA or cardiovascular. The cardiovascular interventions are identified in the vascular surgery database (Karbasen). Major follow-up is performed at 3, 5 and 10 years.

A steering and data validation group will be formed including the project manager and a representative from the Clinical Epidemiology Department. Furthermore, a vascular surgeon from each of the two affected departments in the region will participate.

Total mortality, cardiovascular and AAA-related mortality and initial cardiovascular hospital service are compared for the two groups using Cox proportional hazards-regression analysis which facilitates description of the risk ratio. The cost-efficiency calculation will be adjusted for quality of life.

ELIGIBILITY:
Inclusion Criteria:

* men aged 65-74 years old living in the central region of Denmark

Exclusion Criteria:

* men not aged 65-74 years
* men aged 65-74 years old not living in the central region of Denmark

Ages: 65 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2008-09; Primary Completion 2018-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 3, 5, and 10 years

SECONDARY OUTCOMES:
Cardiovascular events | 3,5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jes S. Lindholt, M.D.,Ph.D., Principal Investigator — Vascular Research Unit, Viborg Hospital
Locations (1):
- Vascular Research Unit, Dept. of Vasc. Surgery, Viborg Hospital, Viborg, Denmark

REFERENCES:
- [Derived] Larsen KL, Kavaliunaite E, Rasmussen LM, Hallas J, Diederichsen A, Steffensen FH, Busk M, Frost L, Urbonaviciene G, Lambrechtsen J, Egstrup K, Lindholt JS. The association between diabetes and abdominal aortic aneurysms in men: results of two Danish screening studies, a systematic review, and a meta-analysis of population-based screening studies. BMC Cardiovasc Disord. 2023 Mar 16;23(1):139. doi: 10.1186/s12872-023-03160-8. PMID 36927295
- [Derived] Lindholt JS, Diederichsen AC, Rasmussen LM, Frost L, Steffensen FH, Lambrechtsen J, Urbonaviciene G, Busk M, Egstrup K, Kristensen KL, Behr Andersen C, Sogaard R. Survival, Prevalence, Progression and Repair of Abdominal Aortic Aneurysms: Results from Three Randomised Controlled Screening Trials Over Three Decades. Clin Epidemiol. 2020 Jan 23;12:95-103. doi: 10.2147/CLEP.S238502. eCollection 2020. PMID 32158272
- [Derived] Lindholt JS, Kristensen KL, Burillo E, Martinez-Lopez D, Calvo C, Ros E, Martin-Ventura JL, Sala-Vila A. Arachidonic Acid, but Not Omega-3 Index, Relates to the Prevalence and Progression of Abdominal Aortic Aneurysm in a Population-Based Study of Danish Men. J Am Heart Assoc. 2018 Jan 26;7(3):e007790. doi: 10.1161/JAHA.117.007790. PMID 29374048
- [Derived] Lindholt JS, Sogaard R. Population screening and intervention for vascular disease in Danish men (VIVA): a randomised controlled trial. Lancet. 2017 Nov 18;390(10109):2256-2265. doi: 10.1016/S0140-6736(17)32250-X. Epub 2017 Aug 28. PMID 28859943
- [Derived] Grondal N, Sogaard R, Henneberg EW, Lindholt JS. The Viborg Vascular (VIVA) screening trial of 65-74 year old men in the central region of Denmark: study protocol. Trials. 2010 May 27;11:67. doi: 10.1186/1745-6215-11-67. PMID 20507582